CLINICAL TRIAL: NCT05466968
Title: Clinical Trial of Suxiao Jiuxin Pill on the Instability of Vulnerable Plaque With Integrated Traditional Chinese Medicine and Western Medicine in Acute ST-segment Elevation Myocardial Infarction(STEMI) Patient
Brief Title: Intervention of Suxiao Jiuxin Pill on Instability of Vulnerable Plaque in Acute Myocardial Infarction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiaolu Li (Other)
Responsible Party: Sponsor-Investigator, Xiaolu Li, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(030)
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; suxiao jiuxin pills

STUDY DESIGN:
Intervention Model Description: Experimental: Suxiao Jiuxin Pills Suxiao Jiuxin Pills prescription (15 pills loading does, maintenance 6 pills each time, three times a day.) for 90 days Placebo Comparator: The placebo of Suxiao Jiuxin Pills The placebo of Suxiao Jiuxin Pills prescription (15 pills loading does, maintenance 6 pills each time, three times a day.) for 90 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drug: Suxiao Jiuxin Pills Suxiao Jiuxin Pills consists Rhizoma Ligustici (Chuan xiong) and Borneolum (Bing pian).
  Drug: The placebo of Suxiao Jiuxin Pills The placebo of Suxiao Jiuxin Pills is similar to Suxiao Jiuxin Pills in appearance, smell, and taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suxiao Jiuxin Pills (Experimental): Suxiao Jiuxin Pills prescription (15 pills loading does, maintenance 6 pills each time, three times a day.) for 90 days
  Interventions: Drug: Suxiao Jiuxin Pills
- The placebo of Suxiao Jiuxin Pills (Placebo Comparator): The placebo of Suxiao Jiuxin Pills prescription (15 pills loading does, maintenance 6 pills each time, three times a day.) for 90 days
  Interventions: Drug: The placebo of Suxiao Jiuxin Pills

INTERVENTIONS:
Drug: Suxiao Jiuxin Pills — Suxiao Jiuxin Pills consists Rhizoma Ligustici (Chuan xiong) and Borneolum (Bing pian).
  Other Names: SJP group
  Arms: Suxiao Jiuxin Pills
Drug: The placebo of Suxiao Jiuxin Pills — The placebo of Suxiao Jiuxin Pills is similar to Suxiao Jiuxin Pills in appearance, smell, and taste.
  Other Names: Con group
  Arms: The placebo of Suxiao Jiuxin Pills

SUMMARY:
The incidence of cardiovascular disease is still high in China under the condition of non-standard treatment of Western medicine. Acute coronary plaque rupture and thrombosis is an extreme manifestation of instability of "vulnerable plaque", which is the result of the joint action of multiple factors. The intervention of unstable plaque reversal from multiple factors is inherently reasonable. Compared with the treatment of thrombosis and unstable plaque in western medicine, quick acting Jiuxin Pill can not only calm and relieve pain for pain and other symptoms, but also regulate immune inflammation and metabolic disorder, improve microcirculation and anti myocardial ischemia. In order to evaluate the efficacy, safety and modern scientific basis of Suxiao Jiuxin Pill in acute myocardial infarction (AMI), the investigators designed this study.

DETAILED DESCRIPTION:
Under the condition of standardized western medicine treatment, the incidence and disability rate of cardiovascular disease in China is still high. There has been a wealth of clinical practice in the treatment of acute myocardial infarction with traditional Chinese medicine, and clinical evidence-based exploration is an inevitable trend. Suxiao Jiuxin Pill is a classic old medicine, but large-scale randomized controlled trial are still needed to consolidate the efficacy, safety and modern scientific basis in acute myocardial infarction (AMI). This pilot single center standardization research is the most basic support and exploration. This project can enhance the influence of Suxiao Jiuxin pills in the context of modern science, which will help the products to be more widely used in Chinese and western hospitals, benefit more patients, reduce the health economics cost of patients with acute ischemia of coronary heart disease at home and abroad, and reduce the social burden. From the perspective of local "vulnerable plaque" instability and "vulnerable patients" systemic inflammation outbreak driving plaque rupture, this study aims to clarify the effect of Suxiao Jiuxin Pill on thrombotic lesions, systemic and clinical short-term prognosis in patients with acute ST segment elevation myocardial infarction (STEMI) from multi-target and multi-component. This study provides evidence for the mechanism of Suxiao Jiuxin Pill in the comprehensive prevention and treatment of pathophysiological disorders in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-75;
2. Meet the diagnosis of AMI global definition version 4，admit from emergency department;
3. Prepare for emergency coronary angiography and PCI reperfusion therapy;
4. Volunteer to participate in this study and have signed an informed consent form.

Exclusion Criteria:

1. AMI with cardiogenic shock (Killip grade ≥ grade III) and no response to vasopressin;
2. AMI complicated with severe arrhythmia (persistent ventricular tachycardia, ventricular fibrillation);
3. AMI complicated with mechanical complications (ventricular septal perforation, papillary muscle rupture, intracardiac thrombus, ventricular free wall rupture);
4. Severe systemic diseases (immune system diseases, sepsis and other serious infections, blood system diseases, massive hemorrhage caused by anticoagulation and antithrombotic therapy, and severe organ failure (such as ALT ≥ 3 ULN, cr> 134 μ Mol/l (2mg/dl) or egfr<45ml/min/1.73m2);
5. History of cerebral hemorrhage and cerebral aneurysm within 3 months;
6. Mental patients;
7. Malignant tumor or other pathophysiological condition with expected survival less than 1 year;
8. Those who are allergic to the drug components of this study;
9. Pregnant or lactating women;
10. Patients who have participated in clinical trials of other drugs within 3 months before enrollment or took other Chinese patent medicines with similar effects within the first three months of enrollment;
11. Other diseases with clinical significance that may cause serious danger to patients.
12. In TCM syndrome types, Qi deficiency, Yang deficiency and other deficiency syndrome types, and cold congealing heart pulse syndrome types in positive syndrome types.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Changes of MMP-9 | Up to 30 minutes after administration
  MMP-9 measure by Elisa

SECONDARY OUTCOMES:
Changes of TIMI myocardial perfusion (TMP) of "criminal vessel". | Up to 30 minutes after administration
  TMP measure by CAG
Changes in the local morphology of vulnerable plaque | Up to 30 minutes after administration
  Proportion of lipid / necrotic core in plaque area by IVUS
Changes of PCSK9 in vulnerable plaque | Up to 30 minutes after administration
  PCSK9 measure by Elisa
Expression changes of local SMC-FC transformation indexes in vulnerable plaque | Up to 30 minutes after administration
  LOX-1 measure by Elisa
Expression changes of Local EC function index of vulnerable plaque | Up to 30 minutes after administration
  iNOS measure by Elisa
Expression changes of Local angiogenic factors in vulnerable plaque | Up to 30 minutes after administration
  VEGF measure by Elisa
Expression changes of indicators associated with vulnerable plaque rupture events | Up to 30 minutes after administration
  TNF-a measure by Elisa
Changes in coagulation related indicators in vulnerable plaque | Up to 30 minutes after administration
  Coagulation factor X measure by Elisa
The changes of inflammation related indicators | 3 months after PCI
  IL-6 by Omics research
Changes of remodeling indexes | 3 months after PCI
  LVEF measure by UCG
Changes in the incidence of MACE | 3 months after PCI
  Recurrent unstable angina pectoris, non fatal myocardial infarction, cardiogenic death, revascularization (pci+cabg), stroke, heart failure requiring hospitalization and all-cause death measure by data statistics

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolu Li, Principal Investigator — Shandong First Medical University
Locations (1):
- Xiaolu Li, Jinan, China